CLINICAL TRIAL: NCT06507878
Title: Global Real World Data in Patients With Advanced Thyroid Cancer on Standard of Care and Specialized Interventions- Registry of Oncologic Outcomes With Testing and Treatment.
Acronym: GRASSROOT
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0394; NCI-2024-06148 (Other: NIH/NCI)
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this clinical research study is to learn about the barriers in the real world to accessing treatments for ATC. And to learn about how patients with ATC tolerate and respond to the commercially available medications for treatment of this disease, outside of a clinical study.

DETAILED DESCRIPTION:
Primary Objectives:

The primary objective of this study is to compare overall survival (OS) between ATC patients treated at MDA versus outside of MDA using treatment regimens offered at MDA based on BRAF status and stage of the disease. We will gather prospective real-world, large-scale, comprehensive data on these patients who are unable to access traditional clinical trials but are treated with MDA regimens, assigned by stage and BRAF-status.

Secondary Objectives:

1. To evaluate effect of chemotherapy, immunotherapy, and radiation therapy on the quality of life for ATC survivors
2. To evaluate how factors such as health insurance and lack of coverage, adherence, and other sociodemographic characteristics influences patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

All adult patients aged 18 years or older with anaplastic thyroid cancer or poorly differentiated thyroid cancer as their clinical and/ or histological diagnosis will be included.

Exclusion Criteria:

Patients who do not have anaplastic thyroid cancer or poorly differentiated thyroid cancer on their tumor tissue would be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 459 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2032-07-01 (Estimated); Study Completion 2034-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Through study completion; an average of 1 year.
  Prospective real-world, large-scale, comprehensive data on these patients who are unable to access traditional clinical trials but are treated with MDA regimens, assigned by stage and BRAF-status.

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka C Iyer, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org